CLINICAL TRIAL: NCT05275400
Title: A Phase 3, Multicenter, Randomized, Parallel-Design, Open-Label Trial to Evaluate the Efficacy and Safety of LY3209590 Compared With Insulin Degludec in Participants With Type 2 Diabetes Currently Treated With Basal Insulin (QWINT-3)
Brief Title: A Study of Insulin Efsitora Alfa (LY3209590) Compared With Insulin Degludec in Participants With Type 2 Diabetes Currently Treated With Basal Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18237; I8H-MC-BDCU (Other: Eli Lilly and Company); 2021-002569-16 (EudraCT Number)
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 500 U/mL - Insulin Efsitora (Experimental): Participants received 500 units per milliliter (U/mL) Insulin Efsitora Alfa (insulin efsitora) administered subcutaneously (SC) once weekly (QW).
  Interventions: Drug: Insulin Efsitora Alfa
- 100 U/mL - Insulin Degludec (Active Comparator): Participants received 100 U/mL insulin degludec administered SC once daily (QD).
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: Insulin Efsitora Alfa — Administered SC
  Other Names: LY3209590 and Basal Insulin-FC
  Arms: 500 U/mL - Insulin Efsitora
Drug: Insulin Degludec — Administered SC
  Arms: 100 U/mL - Insulin Degludec

SUMMARY:
The reason for this study is to see if the study drug insulin efsitora alfa (LY3209590) is safe and effective in participants with Type 2 diabetes that have already been treated with basal insulin. The study consists of a 3-week screening/lead-in period, a 78-week treatment period and a 5-week safety follow-up period. The study will last up to 86 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Type 2 diabetes according to the World Health Organization (WHO) criteria treated with basal insulin
* Are receiving ≥10 units of basal insulin per day and ≤110 units per day at screening
* Have HbA1c value of 6.5% - 10% inclusive, at screening
* Have a Body mass index (BMI) less than or equal to 45 kilogram/square meter (kg/m²)
* Have been treated with one of the following stable insulin regimens at least 90 days prior to screening:

  * once daily U100 or U200 of insulin degludec
  * once daily U100 or U300 of insulin glargine
  * once or twice daily U100 of insulin detemir, or
  * once or twice daily human insulin NPH
* acceptable non insulin glucose lowering therapies may include 0 to up to 3 of the following:

  * dipeptidyl peptidase (DPP-4) IV inhibitors
  * SGLT2 inhibitors
  * metformin
  * alphaglucosidase inhibitors or,
  * Glucagon-Like Peptide-1 (GLP-1) receptor agonists
  * Participants must be willing to stay on stable dose throughout the study

Exclusion Criteria:

* Have Type 1 diabetes mellitus
* Have acute or chronic hepatitis, cirrhosis, or obvious clinical signs or symptoms of any other liver disease, except Nonalcoholic Fatty Liver Disease (NAFLD)
* Estimated glomerular filtration rate (eGFR) <20 milliliters/minute/1.73 square meter (m²)
* Have active or untreated malignancy
* Are pregnant
* Have a significant weight gain or loss the past 3 months
* Have received anytime in the past 6 months, any of the following insulin therapies:

  * prandial insulin
  * insulin mixtures
  * inhaled insulin
  * U-500 insulin, or
  * continuous subcutaneous insulin infusion therapy
* Have had any of New York Heart Association Class IV heart failure or any of the following CV conditions in the past 3 months:

  * acute myocardial infarctions
  * cerebrovascular accident (stroke), or
  * coronary bypass surgery
* Gastrointestinal: have undergone gastric bypass (bariatric) surgery, restrictive bariatric surgery (Lap-Band) or sleeve gastrectomy within 1 year prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (127):
- United States (38):
  - Medical Investigations, Little Rock, Arkansas
  - John Muir Physician Network Research Center, Concord, California
  - AMCR Institute, Escondido, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Diabetes Associates Medical Group, Orange, California
  - University Clinical Investigators, Inc., Tustin, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Encore Medical Research, Hollywood, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Balanced Life Health Care Solutions/SKYCRNG, Lawrenceville, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - L-MARC Research Center, Louisville, Kentucky
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - HealthPartners Institute dba International Diabetes Center, Minneapolis, Minnesota
  - SKY Clinical Research Network Group - Hall, Fayette, Mississippi
  - Clinvest Research LLC, Springfield, Missouri
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - NYC Research, New York, New York
  - Lillestol Research, Fargo, North Dakota
  - Aventiv Research Inc, Columbus, Ohio
  - Intend Research, LLC, Norman, Oklahoma
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Jefferson Clinical Research Institute (JCRI), Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Gadolin Research, Beaumont, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - Juno Research, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (14):
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - Go Centro Medico San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Ciudad Autonoma de Buenos Aire, Buenos Air
  - Stat Research S.A., Ciudad Autónoma de Buenos Aire, Buenos Air
  - Centro Médico Viamonte, Buenos Aires, Ciudad Aut
  - Mautalen Salud e Investigación, Buenos Aires, Ciudad Aut
  - Instituto Centenario, CABA, Ciudad Autónoma de Buenos Aire
  - Centro Medico Privado CEMAIC, Capital, Córdoba Province
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz, Mendoza Province
  - Instituto Médico Catamarca IMEC, Rosario, Santa Fe Province
  - CEMEDIC, Buenos Aires
  - CENUDIAB, Ciudad Autónoma de Buenos Aire
  - Centro Diabetológico Dr. Waitman, Córdoba
- Hungary (6):
  - DRC Gyógyszervizsgáló Központ, Balatonfüred, Veszprém megye
  - Kanizsai Dorottya Korhaz, Nagykanizsa, Zala County
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg, Zala County
  - Szent Margit Rendelointézet, Budapest
  - Szent János Kórház, Budapest
  - Strazsahegy Medicina Bt., Budapest
- Japan (20):
  - Tokuyama Clinic, Mihama-ku,Chiba City, Chiba
  - Yuri Ono Clinic, Sapporo, Hokkaido
  - Nakamoto Internal Medicine Clinic, Mito, Ibaraki
  - Kozawa Eye Hospital and Diabetes Center, Mito, Ibaraki
  - Noritake Clinic, Ushiku, Ibaraki
  - Matoba Internal Medicine Clinic, Ebina, Kanagawa
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi, Kanagawa
  - Shiraiwa Medical Clinic, Kashihara, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Shimizu Clinic Fusa, Saitama-shi, Saitama
  - Oyama East Clinic, Oyama, Tochigi
  - Tokyo-Eki Center-building Clinic, Chuo Ku, Tokyo
  - The Institute of Medical Science, Asahi Life Foundation, Chuo-ku, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Jinnouchi Hospital, Kumamoto
  - Heiwadai Hospital, Miyazaki
  - AMC Nishiumeda Clinic, Osaka
  - Abe Clinic, Ōita
- Poland (11):
  - OMEDICA Medical Center, Poznan, Greater Poland Voivodeship
  - Gaja Poradnie Lekarskie Maciej Wiza, Poznan, Greater Poland Voivodeship
  - NZOZ Diab-Endo-Met, Krakow, Lesser Poland Voivodeship
  - Private Practice - Dr. Robert Witek, Tarnów, Lesser Poland Voivodeship
  - CenterMed Lublin NZOZ, Lublin, Lublin Voivodeship
  - Gabinety TERPA, Lublin, Lublin Voivodeship
  - NZOZ Medica, Lublin, Lublin Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska, Silesian Voivodeship
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
  - IRMED, Piotrkow Trybunalski, Łódź Voivodeship
- Puerto Rico (2):
  - GCM Medical Group, PSC - Hato Rey Site, San Juan, PR
  - Mgcendo Llc, San Juan
- Slovakia (7):
  - MediVet s.r.o., Malacky, Bratislava Region
  - Human Care s.r.o., Košice, Košice Region
  - Areteus s.r.o., Trebišov, Košice Region
  - MEDI-DIA s.r.o., Sabinov, Presov
  - Diacrin .s.ro., Bratislava
  - DIA-MED CENTRUM s.r.o., Púchov
  - ENDIAMED s.r.o, Dolný Kubín, Žilina Region
- South Korea (12):
  - Kangwon National University Hospital, Chuncheon, Kang-won-do
  - Yonsei University-Wonju Severance Christian Hospital, Wŏnju, Kang-won-do
  - Korea University Ansan Hospital, Ansan-si, Kyǒnggi-do
  - Hanyang University Guri Hospital, Guri-si, Kyǒnggi-do
  - Yeungnam Univeristy Medical Center, Gyeongsan-si, Kyǒngsangbuk-do
  - Inje University Sanggye Paik Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Hallym University Kangnam Sacred Heart Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kyung Hee University Hospital at Gangdong, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teuk
  - Ulsan University Hospital, Ulsan, Ulsan-Kwangyǒkshi
- Spain (11):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [La Coruña]
  - Centro Periférico de Especialidades Bola Azul, Almería, Almería
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Quiron Infanta Luisa, Seville, Andalusia
  - Clínica Juaneda, Palma de Mallorca, Balears [Baleares]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Vithas Hospital Sevilla, Seville, Sevilla
  - Hospital Universitario de La Ribera, Alzira, Valenciana, Comunitat
  - Hospital General Universitario de Valencia, Valencia, Valenciana, Comunitat
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
- Taiwan (6):
  - Chung Shan Medical University Hospital, Taichung, Taichung
  - Taichung Veterans General Hospital, Taichung, Taichung
  - Chi Mei Medical Center, Tainan, Tainan
  - Fu Jen Catholic University Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Miller E, Davidson MB, Bajaj HS, Rosenstock J, Philis-Tsimikis A, Bergenstal RM, Case M, Ilag L, Threlkeld R, Levasseur E, Gelsey F. Evaluation of Overall Health State, Treatment Burden, and Satisfaction with Insulin Efsitora Alfa (Efsitora) vs. Daily Comparator in Adults with Type 2 Diabetes in the QWINT Clinical Trial Program. Diabetes Ther. 2026 Jan 27. doi: 10.1007/s13300-025-01833-5. Online ahead of print. PMID 41591636
- [Derived] Philis-Tsimikas A, Bergenstal RM, Bailey TS, Jinnouchi H, Thrasher JR, Ilag L, Mitra J, Syring K, Threlkeld RJ. Once-weekly insulin efsitora alfa versus once-daily insulin degludec in adults with type 2 diabetes currently treated with basal insulin (QWINT-3): a phase 3, randomised, non-inferiority trial. Lancet. 2025 Jun 28;405(10497):2279-2289. doi: 10.1016/S0140-6736(25)01044-X. Epub 2025 Jun 22. PMID 40562047
- See also: A Study of LY3209590 Compared With Insulin Degludec in Participants With Type 2 Diabetes Currently Treated With Basal Insulin — https://trials.lillytrialguide.com/en-US/trial/2r9JxzEnerVifDDkc8VETS

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants underwent a 3 week screening and lead-in period, and a 78-week treatment period, followed by a 5-week safety follow-up period.
Period: Treatment Period
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Started | 655 | 331
Received At Least 1 Dose of Study Drug | 655 | 331
Completed | 593 | 303
Not Completed | 62 | 28
Not completed — Adverse Event | 7 | 1
Not completed — Assigned Treatment by Mistake | 6 | 3
Not completed — Death | 5 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 5 | 4
Not completed — Non-Compliance with Study Drug | 5 | 1
Not completed — Withdrawal by Subject | 30 | 12
Not completed — Lost to Follow-up | 1 | 5
Not completed — Lack of Efficacy | 1 | 0
Not completed — Sponsor Decision | 1 | 0
Period: Follow-Up Period
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Started | 614 (Per protocol, participants who completed the study treatment period were required to complete a safety follow-up period and participants who discontinued the study treatment prematurely were encouraged to remain in the study for safety monitoring.) | 306 (Per protocol, participants who completed the study treatment period were required to complete a safety follow-up period and participants who discontinued the study treatment prematurely were encouraged to remain in the study for safety monitoring.)
Completed | 608 | 306
Not Completed | 6 | 0
Not completed — Death | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- 500 U/mL - Insulin Efsitora: Participants received 500 U/mL insulin efsitora administered SC QW.
- 100 U/mL - Insulin Degludec: Participants received 100 U/mL insulin degludec administered SC QD.
- Total: Total of all reporting groups
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec | Total
Number analyzed (Participants) | 655 | 331 | 986
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.60 (10.17) | 60.80 (9.97) | 60.70 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 279 | 152 | 431
  Male | 376 | 179 | 555
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 179 | 88 | 267
  Not Hispanic or Latino | 476 | 243 | 719
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 180 | 92 | 272
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 32 | 20 | 52
  White | 438 | 218 | 656
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 103 | 52 | 155
  Hungary | 24 | 14 | 38
  Japan | 94 | 47 | 141
  Poland | 59 | 29 | 88
  Slovakia | 60 | 31 | 91
  South Korea | 64 | 31 | 95
  Spain | 52 | 25 | 77
  Taiwan | 19 | 11 | 30
  United States | 180 | 91 | 271
HemoglobinA1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 7.8 (0.9) | 7.8 (0.9) | 7.8 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) [Noninferiority]
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) Mean was determined using ANCOVA model with Baseline + Country + Type of Basal Insulin used at Baseline + Treatment (Type III sum of squares) as variables. Missing data at Week 26 were imputed by return-to-baseline multiple imputation approach.
Time Frame: Baseline, Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome at baseline or week 26. Participants who were assigned treatment by mistake were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 649 | 328
Percentage of HbA1c | -0.81 (0.0302) | -0.72 (0.0424)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Non-Inferiority — Noninferiority margin (NIM) was 0.4%; LS Mean Difference = -0.089, 95% CI 2-sided [-0.191 to 0.013]

2. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) [Superiority]
Description: as for outcome 1
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 649 | 328
Percentage of HbA1c | -0.81 (0.0302) | -0.72 (0.0424)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.088, ANCOVA; LS Mean Difference = -0.089, 95% CI 2-sided [-0.191 to 0.013]

3. Secondary Outcome: Nocturnal Hypoglycemia Event Rate
Description: The event rate of participant-reported clinically significant glucose <54 mg/dL (3.0 mmol/L) or severe nocturnal hypoglycemia that occurs at night and presumably during sleep between midnight and 6:00 AM), measured during treatment period up to week 78. Group mean is reported here. Group mean is determined by Negative Binomial Model using Number of episodes = Hemoglobin A1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline up to Week 78
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Error); unit: Events per year
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 655 | 331
Events per year | 0.11 (0.022) | 0.10 (0.019)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.897, Negative binomial model; Relative rate = 1.03, 95% CI 2-sided [0.62 to 1.74]

4. Secondary Outcome: Percentage of Time in Glucose Range Between 70 and 180 mg/dL (3.9 and 10.0 mmol/L)
Description: Percentage of time in glucose range between 70 and 180 mg/dL (3.9 and 10.0 millimoles per liter (mmol/L)) inclusive measured by continued glucose monitoring (CGM) during CGM session prior to week 26. LS Mean was calculated using ANCOVA model with Baseline + Country + Hemoglobin A1c Stratum at Baseline + Type of Basal Insulin used at Baseline + Treatment (Type III sum of squares) as variables. Missing data during CGM session prior to Week 26 were imputed by return-to-baseline multiple imputation approach.
Time Frame: Week 22 to Week 26
Population: All randomized participants who took at least one dose of the study drug and had evaluable data for this outcome at baseline or Week 22-26 were included. Participants who were assigned treatment by mistake were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 641 | 325
Percentage of time | 61.37 (0.676) | 60.95 (0.954)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.722, ANCOVA; LS Mean Difference = 0.42, 95% CI 2-sided [-1.88 to 2.72]

5. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Fasting glucose measured by Self-Monitoring of Blood Glucose (SMBG). LS Mean was determined using ANCOVA model with Baseline + Country + Type of Basal Insulin at Baseline + Baseline HbA1C Stratum (%) + Treatment (Type III sum of squares) as variables. Missing data at baseline are imputed with multiple imputation under assumption of missing at random. Missing data at Week 26 are imputed by return-to-baseline multiple imputation approach.
Time Frame: Baseline, Week 26
Population: All randomized participants who took at least one dose of the study drug and had evaluable data for this outcome at baseline or Week 26 were included. Participants who were assigned treatment by mistake were excluded.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 648 | 327
milligrams per deciliter (mg/dL) | -30.97 (0.943) | -30.13 (1.323)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.605, ANCOVA; LS Mean Difference = -0.84, 95% CI 2-sided [-4.01 to 2.33]

6. Secondary Outcome: Weekly Insulin Dose at Week 26
Description: The average weekly insulin dose at Week 26 was reported. LS Mean was determined by mixed model repeated measures (MMRM) model using BASELINE + Country + Type of Basal Insulin at Baseline + Baseline HbA1C Stratum (%) + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-covariance structure was set as compound symmetry.
Time Frame: Week 26
Population: All participants who received at least one dose of study drug, had a baseline and at least one post-baseline value for this outcome. Participants who were assigned treatment by mistake were excluded.
Measure: Least Squares Mean (Standard Error); unit: Units per week of insulin
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 647 | 327
Units per week of insulin | 333.20 (5.93) | 363.20 (8.33)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.003, Mixed Models Analysis; LS Mean Difference = -30.00, 95% CI 2-sided [-50.10 to -9.97]

7. Secondary Outcome: Hypoglycemia Event Rate
Description: Patient reported events of hypoglycemia - Hypoglycemia with glucose <54 mg/dL (Level 2) or Severe Hypoglycemia (Level 3) was reported. A severe hypoglycemic event is characterized by altered mental or physical status requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions for the treatment of hypoglycemia. Group mean was reported and determined by Negative binomial method using Hemoglobin A1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as variables.
Time Frame: Baseline up to Week 78
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Error); unit: Events per year
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 655 | 331
Events per year | 0.84 (0.082) | 0.74 (0.098)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.430, Negative binomial model; Relative rate = 1.14, 95% CI 2-sided [0.83 to 1.56]

8. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was reported. LS Mean was determined by MMRM model using BASELINE + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 78
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 654 | 330
kilograms (kg) | 2.27 (0.133) | 2.20 (0.186)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.756, Mixed Models Analysis; LS Mean Difference = 0.071, 95% CI 2-sided [-0.38 to 0.52]

9. Secondary Outcome: Percentage of Time in Hypoglycemia Range
Description: Percentage of time in hypoglycemia range with glucose <54 mg/dL (3.0 mmol/L) measured during CGM from 22-26 weeks. LS Mean was determined using ANCOVA model using Baseline + Country + Hemoglobin A1c Stratum at Baseline + Type of Basal Insulin used at Baseline + Treatment (Type III sum of squares) as variables. Missing data at baseline were imputed with multiple imputation under assumption of missing at random. Missing data at Week 22-26 were imputed by return-to-baseline multiple imputation approach.
Time Frame: Week 22 to Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 641 | 325
Percentage of time | 0.36 (0.036) | 0.22 (0.051)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.021, ANCOVA; LS Mean Difference = 0.14, 95% CI 2-sided [0.02 to 0.27]

10. Secondary Outcome: Percentage of Time in Hyperglycemia Range
Description: Percentage of time in hyperglycemia range with glucose >180 mg/dL (10.0 mmol/L) measured during the CGM session from 22-26 weeks. LS Mean was determined using ANCOVA model using Baseline + Country + Hemoglobin A1c Stratum at Baseline + Type of Basal Insulin used at Baseline + Treatment (Type III sum of squares) as variables. Missing data at baseline were imputed with multiple imputation under assumption of missing at random. Missing data at Week 22-26 were imputed by return-to-baseline multiple imputation approach.
Time Frame: Week 22 to Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 641 | 325
Percentage of time | 37.25 (0.700) | 38.24 (0.989)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.417, ANCOVA; LS Mean Difference = -0.99, 95% CI 2-sided [-3.37 to 1.40]

11. Secondary Outcome: Change From Baseline in Treatment-Related Impact Measure - Diabetes (TRIM-D)
Description: The TRIM-D is a self-administered instrument, which assesses the impact of diabetes treatment on participants' functioning and well-being across available diabetes treatments. The TRIM-D consists of 28 items each assessed on a 5-point scale. TRIM-D items assess 5 domains of impact:
  * Treatment Burden (6 items)
  * Daily Life (5 items)
  * Diabetes Management (5 items)
  * Compliance (4 items), and
  * Psychological Health (8 items)
  Items within each domain are summed to obtain a raw domain score, which is then transformed to a 0-100 scale, where higher scores indicate a greater impact on participant's functioning and well-being.
  LS mean was determined using MMRM model with BASELINE + Country + Type of Basal Insulin at Baseline + Baseline HbA1C Stratum (%) + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: All participants who received at least one dose of the study drug, had a baseline and at least one post-baseline value for this outcome. Participants who were assigned treatment by mistake were excluded.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 625 | 314
Score on a scale
  Week 26 | 10.03 (0.424) | 6.88 (0.599)
  Week 52: number analyzed (Participants) | 580 | 294
  Week 52 | 10.09 (0.445) | 6.53 (0.627)
  Week 78: number analyzed (Participants) | 548 | 281
  Week 78 | 10.33 (0.472) | 6.98 (0.662)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Week 26; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 3.15, 95% CI 2-sided [1.71 to 4.59]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Week 52; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 3.56, 95% CI 2-sided [2.05 to 5.07]
Statistical Analysis 3: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Degludec; Week 78; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 3.35, 95% CI 2-sided [1.75 to 4.94]

12. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire-Change Version (DTSQc) - Treatment Satisfaction Score: Week 26
Description: DTSQc treatment satisfaction score is a 6-item questionnaire which assesses relative change in overall treatment satisfaction. The treatment satisfaction score ranges from -18 to 18, where higher the score the greater the improvement in satisfaction with treatment. The lower the score the greater the deterioration in satisfaction with treatment.
Time Frame: Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome. Participants who were assigned treatment by mistake were excluded.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 599 | 304
Score on a scale | 14.9 (4.47) | 12.3 (6.15)

13. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire-Change Version (DTSQc) - Treatment Satisfaction Score: Week 52
Description: as for outcome 12
Time Frame: Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 570 | 290
Score on a scale | 15.1 (4.45) | 12.3 (6.10)

14. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire-Change Version (DTSQc) - Treatment Satisfaction Score: Week 78
Description: as for outcome 12
Time Frame: Week 78
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 523 | 268
Score on a scale | 15.4 (4.23) | 11.7 (6.61)

ADVERSE EVENTS:
Time Frame: Baseline Through Safety Follow-Up (Up to 83 Weeks)
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 7/655 | 2/331
Serious Adverse Events (participants affected / at risk) | 103/655 | 37/331
Other Adverse Events (participants affected / at risk) | 241/655 | 102/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 500 U/mL - Insulin Efsitora (N=655) | 100 U/mL - Insulin Degludec (N=331)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 4 (4)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 5 (5) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 4 (4)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1/376 (1) | 0/179 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Primary hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 3 (3) | 1 (1)
Diabetic retinopathy (Eye disorders) | 2 (2) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 2 (2) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Acute cholecystitis necrotic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hcov-oc43 infection (Infections and infestations) | 1 (1) | 0 (0)
Hiv infection (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of asthma (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (3) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Continuous glucose monitoring (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/279 (0) | 1/152 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/376 (4) | 0/179 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dural arteriovenous fistula (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/376 (1) | 0/179 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 2 (2) | 0 (0)
Limb amputation (Surgical and medical procedures) | 1 (2) | 0 (0)
Skin graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Aneurysm thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 2 (3) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500 U/mL - Insulin Efsitora (N=655) | 100 U/mL - Insulin Degludec (N=331)
Diarrhoea (Gastrointestinal disorders) | 35 (46) | 14 (23)
Covid-19 (Infections and infestations) | 70 (73) | 27 (28)
Nasopharyngitis (Infections and infestations) | 60 (88) | 29 (36)
Upper respiratory tract infection (Infections and infestations) | 34 (40) | 18 (25)
Dose calculation error (Injury, poisoning and procedural complications) | 42 (55) | 15 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (39) | 12 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (35) | 12 (12)
Headache (Nervous system disorders) | 36 (57) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT05275400/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT05275400/SAP_001.pdf